CLINICAL TRIAL: NCT04304729
Title: Early Myocardial Morphologic and Functional Changes and Their Association With Diet and Physical Activity in Adolescents With Type 1 Diabetes
Brief Title: Determinants of Cardiovascular Disease Risk Factors Among Youth With Type 1 Diabetes
Acronym: CARDEA
Status: Suspended | Type: Observational
Why Stopped: Recruitment for phase 1 is completed, waiting for phase 2
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Melanie Henderson, Associate professor, Pediatrics, St. Justine's Hospital
Other Study IDs: 2016-936; 366194 (Other Grant/Funding Number: Canadian Institutes of Health Research); G-16-00012590 (Other Grant/Funding Number: Heart and Stroke Foundation of Canada)
Record Dates: First submitted 2020-02-27; First posted 2020-03-11 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes; Cardiovascular Risk Factor
Keywords: Type 1 Diabetes; Cardiovascular disease; Adolescents; Cardiac MRI; Diet; Physical activity; Sedentary behavior; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, whole blood, urine, feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics: Girls and boys living with Type 1 Diabetes.
- Control: Age and sex matched participants without any type of diabetes

SUMMARY:
Type 1 diabetes mellitus (T1D) is the most common form of diabetes among children and youth, and it is increasing around the world, particularly among children under 5 years. This is worrisome given the chronic nature of the disease and its strong association with an increased risk of cardiovascular disease (CVD). Evidence suggests that markers of CVD are already present in children with T1D, making prevention a clinical and public health priority in this high-risk population. Despite this, a good understanding of what factors predispose children with T1D to CVD is still lacking.

Our study aims to better understand in this population what individual, familial and environmental characteristics increase the risk for heart disease, how to best measure it early on and what are the potential mechanisms underlying the heightened risk for heart disease in youth with T1D. Specifically, we aim to:

1. compare established risk factors (dyslipidemia, hypertension) with novel early markers for CVD (cardiac phenotype, arterial stiffness, endothelial function) in adolescents with T1D and healthy controls;
2. examine the associations between these novel early markers with: i) lifestyle habits; ii) measures of inflammation; and iii) markers of oxidative stress among adolescents with T1D and healthy controls, and determine group differences in these associations;
3. explore, across both groups, the associations between these established and novel early markers of CVD with neighborhood features.
4. Determine sex and gender differences in novel markers of CVD (cardiac structure/myocardial oxygenation, vascular studies including endothelial function and arterial stiffness) in youth with T1D and healthy controls;
5. Determine, across both groups, sex and gender differences in associations between markers of CVD and lifestyle habits, specifically: i) moderate-to-vigorous physical activity (MVPA); ii) dietary intake (carbohydrates, sugar, saturated/trans-fat, fiber, food groups); iii) sedentary behavior; and iv) sleep;
6. Measure changes in novel markers of CVD from adolescence to early adulthood among individuals with T1D and healthy controls;
7. Assess whether lifestyle habits in adolescence are prospectively associated with established (dyslipidemia, hypertension) and novel (cardiac structure/myocardial oxygenation, endothelial function, arterial stiffness) markers of CVD in early adulthood, and if these associations differ according to T1D status, adiposity, sex and gender.

To achieve these objectives, we will compare 300 participants aged 14-18 years with T1D to 300 healthy controls. 100 participants from each group will be reassessed at the age of 22-26 yo. Lifestyle habits include assessments of physical activity, sleep, sedentary behavior, fitness and dietary intake. Blood pressure and lipid profiles will be measured. Cardiac structure/function will be evaluated by non-contrast cardiac magnetic resonance imaging (CMR). Aortic distensibility will be determined by pulse wave velocity. Endothelial function will be determined by flow-mediated dilation. Inflammatory markers and endogenous antioxidants will be measured in blood. Intestinal microbiota will be assessed. Neighbourhood features include built and social environment indicators and air quality.

Our study provides an exceptional opportunity to increase our knowledge on what factors predispose children with T1D to cardiovascular disease. Understanding the interplay between T1D, lifestyle habits and metabolic markers and CVD is critical to developing effective prevention strategies for these vulnerable children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D (for the T1D group) or no diagnosis of any type of diabetes (for the control group)
* 14 to 18 years old

Exclusion Criteria:

* Youth with another type of diabetes such as T2D
* Conditions that could limit their ability to participate in the study
* Known pathology that would influence their risk for CVD
* Siblings of a participant already enrolled in the study

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: T1D group: Sainte-Justine Hospital's Diabetes Clinic patients
  Control group: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac structure (MRI) | Baseline measurement
Endothelial function (Flow-mediated dilation) | Baseline measurement
Vascular structure (Pulse-wave velocity) | Baseline measurement

SECONDARY OUTCOMES:
Dyslipidemia | Baseline measurement
Hypertension | Baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Henderson, MD, Ph.D, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Henderson M, Friedrich M, Van Hulst A, Pelletier C, Barnett TA, Benedetti A, Bigras JL, Drapeau V, Lavoie JC, Levy E, Mathieu ME, Nuyt AM. CARDEA study protocol: investigating early markers of cardiovascular disease and their association with lifestyle habits, inflammation and oxidative stress in adolescence using a cross-sectional comparison of adolescents with type 1 diabetes and healthy controls. BMJ Open. 2021 Sep 8;11(9):e046585. doi: 10.1136/bmjopen-2020-046585. PMID 34497076